CLINICAL TRIAL: NCT03686410
Title: Effects of a Web-based Therapeutic Educational Intervention About Pain and Poor Sleep Quality in Women Diagnosed With Fibromyalgia: a Mixed Methods Research With Sequential Exploratory Design
Brief Title: Therapeutic Educational Intervention and Fibromyalgia: a Mixed Methods Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Carolina Climent-Sanz, Pre-doctoral fellow, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULeida
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Therapeutic Patient Education; Educational Technology; Mixed Methods Research; Pain; Poor Sleep Quality
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the participants and the study researchers will not know the group assigned to each subject. In fact, the evaluations will be carried out through the website.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Therapeutic Educational Intervention (Experimental): The subjects assigned to this group will follow a web-based therapeutic educational intervention on pain and poor sleep quality.
  All the subjects assigned to this intervention will have free access to the website from any device with internet access and will be able to consult it as many times as they wish during the intervention. The intervention will last for four weeks.
  Interventions: Behavioral: Web-based Therapeutic Educational Intervention
- 2. Convetional Tretament (Active Comparator): The subjects assigned to this condition will continue with their usual treatment is based on the recommendations of the clinical practice guideline for the treatment of fibromyalgia "Guide of Fibromyalgia" developed by the Department of Health of the Generalitat de Catalunya and the Servei Català de Salut.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Behavioral: Web-based Therapeutic Educational Intervention — The subjects assigned to this group will follow a web-based therapeutic educational intervention on pain and poor sleep quality.
  All the subjects assigned to this intervention will have free access to the website from any device with internet access and will be able to consult it as many times as they wish during the intervention. The intervention will last for four weeks.
  Arms: 1. Therapeutic Educational Intervention
Other: Conventional Treatment — The subjects assigned to this condition will continue with their usual treatment is based on the recommendations of the clinical practice guideline for the treatment of fibromyalgia "Guide of Fibromyalgia" developed by the Department of Health of the Generalitat de Catalunya and the Servei Català de Salut.
  Arms: 2. Convetional Tretament

SUMMARY:
Fibromyalgia is the most common central sensitivity syndrome and one of the principal causes of chronic widespread pain among the adult population worldwide. Recent studies indicated that poor sleep quality is highly prevalent and a troublesome symptom among patients with fibromyalgia. Psychosocial and behavioral factors have been demonstrated to be intimately related with the symptomatic experience of fibromyalgia patients. Pain catastrophizing and dysfunctional beliefs and attitudes about sleep are involved in the perpetuation of those symptoms and affecting other spheres of the syndrome Objective: The aim of this project is to evaluate the cognitive and behavioral factors related with pain and poor sleep quality in women diagnosed with fibromyalgia so as to develop and test the effects of a web-based therapeutic educational intervention about pain and sleep on pain intensity, pain catastrophizing, sleep quality, dysfunctional beliefs and attitudes about sleep, and quality of life and health status related with fibromyalgia Methods: A mixed methods research with sequential exploratory design will be applied. For the qualitative phase, a snowballing sampling technique will be used. The participants will be invited to participate in a personal semi-structured interview. For the quantitative phase a sample of 64 adult women with fibromyalgia will be recruited from primary care centers of the city of Lleida and randomized into either the intervention or the control group Discussion: There is an imperative necessity of taking patients' symptoms experience as essential for the development of effective symptom management strategies from a biopsychosocial perspective. In the era of the internet, our web-based therapeutic educational intervention could open a new window for the treatment of women with fibromyalgia as part of current FM management treatments in primary care.

Our hypotheses are:

* Cognitive and behavioral factors related to pain and poor sleep quality in women diagnosed with fibromyalgia act as perpetuating factors and aggravate the general health status and the quality of life of these patients.
* A web-based therapeutic educational intervention about pain and poor sleep quality in women diagnosed with FM is better than the conventional approach for the treatment of pain intensity, pain catastrophizing, sleep quality, dysfunctional beliefs and attitudes about sleep, and general health status and quality of life-related with FM.

DETAILED DESCRIPTION:
Study design Mixed method research with a sequential exploratory design.

A three-stage procedure will be used:

1. Qualitative phase: collection and analysis of qualitative data.
2. Connection phase: based on the results obtained in the previous stage the content of the educational intervention will be developed.
3. Quantitative phase: the resulting educational intervention will be tested in a sample of the target population and subsequently the quantitative data will be collected and analyzed.

Qualitative Phase Objective To explore the evaluation (cognitive factors) and response (behavioral factors) associated with pain and poor sleep quality in Spanish women diagnosed with Fibromyalgia.

Methodological orientation and Theory Generic qualitative study Sampling, Sample Size, and Method of Approach In this phase, a non-probabilistic snowball sampling technique will be used. The inclusion of participants will stop when new ideas or data about the research topic stop appearing, that is, until the information is saturated.

Women who agree to participate in the qualitative phase will be contacted by the principal investigator to assess compliance with the established inclusion criteria and to read and sign the informed consent.

Data collection and analysis Qualitative data will be collected through in-depth semi-structured individual interviews.

The interviews will be conducted individually by the main researcher of the study in Spanish or Catalan, depending on the mother tongue of the interviewee. Also, the interview will be held in a place chosen by the participants to facilitate a comfortable environment.

All interviews will be recorded in digital format, transcribed and subsequently imported into the qualitative analysis software ATLAS.ti. A triangulation of researchers will be conducted.

Connection Phase The connection phase is of special importance in the development of projects with exploratory sequential mixed methodology since it is in this phase where the integration of the qualitative and quantitative phases is clear. In this project, the data of the qualitative phase are essential for the development of the content of the therapeutic educational intervention, whose effects will be evaluated in the quantitative phase by means of an RCT.

Once the qualitative data is analyzed the author will develop the content of the therapeutic educational intervention and the materials (videos, dossiers) that will be available on the website for the participants of the study.

Using the data of the qualitative phase for the development of the therapeutic educational intervention will assure that the materials are based on the FM patients' needs. The best and most current scientific evidence will be consulted so as to provide the participants with a high-quality website with proper information about pain and sleep in the context of FM. The latter is what makes this project an innovative approach in this field of research aimed to respond to the actual needs of FM patients' based on their own experience.

With the help of an information technology technician, the author will design, create and maintain the website. The website will be only accessible with a user number and password provided by the author to the participants once they are allocated to the treatment conditions.

Quantitative Phase Hypothesis A web-based therapeutic educational intervention on pain and poor sleep quality shows more significant clinical effects than the conventional medical treatment for the management of pain, poor sleep quality, catastrophizing of pain, beliefs and dysfunctional attitudes in relation to sleep and the state of health and quality of life associated with fibromyalgia in Spanish women diagnosed with fibromyalgia in a primary care setting.

Principal Objective To evaluate the effects of a web-based therapeutic educational intervention on pain intensity and sleep quality in Spanish women diagnosed with fibromyalgia compared to conventional treatment.

Secondary Objectives

To evaluate the effects of a web-based therapeutic educational intervention in Spanish women diagnosed with fibromyalgia compared to conventional treatment on:

* Pain Catastrophizing
* Dysfunctional beliefs and attitudes in relation to sleep
* Health status, functionality, and quality of life associated with FM Study Design A parallel, double-blind randomized controlled trial. Setting of the study Primary care centers in the city of Lleida Recruitment and sampling method Patients will be recruited from the Primary Care Centers of the city of Lleida. A list of women diagnosed with fibromyalgia will be requested to the board of the primary care of the city of Lleida.

A systematized sampling method will be used in order to assure that all the women in the list have the same chance for participating in the study. The principal investigator will call the women on the list and will meet whit those showing interest in participating so as to assess compliance with the inclusion criteria and to provide them with the information sheet and informed consent.

Intervention plan Experimental group: the subjects assigned to this group will follow a web-based therapeutic educational intervention about pain and poor sleep quality.

All the subjects assigned to this intervention will have free access to the website from any device with internet access and will be able to consult it as many times as they wish during the intervention.

Control group: the subjects assigned to this condition will continue with their usual treatment is based on the recommendations of the clinical practice guidelines for the treatment of FM "Guide of Fibromyalgia" developed by the Department of Health of the Generalitat de Catalunya and the Servei Català de Salut.

Outcomes Primary outcomes

* Pain intensity
* Sleep Quality
* Pain Catastrophizing
* Dysfunctional Beliefs and Attitudes about Sleep
* Health status and quality of life associated with fibromyalgia:

Sample Size According to the Granmo sample size calculation program, accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 32 subjects are required in the first group and 32 in the second to detect a difference equal to or greater than 15 units. It is assumed that the common standard deviation is 12.63. A tracking loss rate of 20% has been estimated.

Randomization Type and Sequence Generation A simple randomization method will be used. A 1:1 ratio will be established for the allocation of participants in each group so that there is the same number of subjects in the experimental and in the control group. The randomization list will be generated through the STATS® computer program by a person specializing in statistics and not related to the study.

Allocation Concealment Mechanism and Implementation In order not to infer in a selection bias, the allocation must be hidden from the researchers responsible for the recruitment of patients. In the case of the present investigation, and given that the pertinent evaluations will be made through the website, there will be no researchers in charge of assessing the participants.

To ensure allocation concealment, a centralized randomization will be carried out through the internet. When the principal researcher ensures compliance with the inclusion criteria and the participant reads, accepts and signs the informed consent, the participants' number will be requested online. This number will not be in any way related to the intervention groups, so neither the researcher nor the participant can anticipate their assignment.

This same number will be entered on the website by the patient when she accesses the website and at that moment she will know the instructions to follow on the screen according to the group to which she has been assigned.

Blinding A double-blind study is proposed in which the participants and the study researchers will not know the group assigned to each subject. In fact, the evaluations will be carried out through the website.

Data Collection The variables to be studied will be evaluated through the questionnaires previously presented which must be completed by the participants of both intervention groups through the website at pre and post-intervention and at three and six months after the intervention.

In each of these five moments of data collection, the subjects of both treatment conditions will receive an email and WhatsApp as a reminder when the questionnaires are available in the website, if they still do not complete the questionnaires, they will be contacted by telephone.

The questionnaires of each patient will be automatically sent to a database to which only the statistician will have access. After each assessment moment, the data obtained will be exported to the "Statistical Package for Social Sciences Software" (SPSS).

Statistical Analysis For the univariate analysis, the variables will be described through measures of central tendency and position, such as the mean, the median, and the mode; dispersion measures such as interquartile range, standard deviation and variance. They will be represented by graphs and tables in order to facilitate the reading of the data.

Regarding the bivariate analysis, the Chi2 statistical coefficient of Pearson and the t-Student test will be used to determine whether or not there is a relationship between the dependent variables and the independent variables.

The statistical analysis to determine the statistical significance will be carried out assuming a confidence interval of 95% and an alpha value of 5% (0.05).

In relation to the clinical significance, the following values will be established:

* Pain intensity (VAS): it is established that a decrease of between 10 and 20% of pain intensity as the minimum clinically important difference, a change of ≥30% as a moderate clinical difference and, finally, a reduction in pain intensity ≥50% reflects substantial changes (32).
* Pain Catastrophizing (PCS): a reduction of the 15-30% is established as the minimum clinically significant change, changes between 30 and 50% are moderately clinically significant and reductions of ≥50% are indicative of substantial clinical improvement (37).
* Health status and Quality of Life related with FM (FIQ-R): a 45.5% change or a change of 27.04 points in the total score of the FIQ is established as the minimum clinically meaningful change (46).
* For the measurement tools whose minimal clinically important difference has not yet been determined, the Standard Median Deviation will be calculated.

ETHICAL ISSUES This study follows the basic ethical principles of respect for people, beneficence and justice established in the Belmont Report, the moral, ethical and legal principles of the Nuremberg Code, the principles of medical research that include human subjects of the Declaration of Helsinki and the "Guideline for Good Clinical Practice" (CPMP/ICH/135/95).

Also, given the management and use of personal data of the participants in both phases of the project and the use of a website for the development of the therapeutic educational intervention, this research will be subject to the "Reglamento (UE) 2016/679 del Parlamento Europeo y del Consejo de 27 de abril de 2016 relativo a la protección de las personas física en lo que respecta al tratamiento de datos personales y a la libre circulación de estos datos".

All participants will be provided with an informed consent document that will be accompanied by a full explanation regarding the investigation, the use of the data by the authors, as well as the laws that protect their rights.

As the intervention does not involve any physical activity/intervention, we expect not to have any physical side effect. However, patients will be advised to contact their family physician if they have any physical problem or any worsening of their condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia based on the 2016 criteria of the American College of Rheumatology
* Women in adulthood: between 18 and 65 years of age
* Understand and speak Spanish and/or Catalan
* Accept and sign the informed consent

Exclusion Criteria:

* Be receiving or having received interventions similar to this study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  Visual Analogue Scale: It was developed in the second half of the seventies and is considered the most sensitive test for the measurement of pain intensity. It is a user-friendly tool which consists of a numerically graduated line from 0-100, with 0 "no pain" and 100 "unbearable pain". Based on the research of Dworkin et al. it is established that a decrease of between 10 and 20% of pain intensity as the minimum clinically important difference, a change of ≥30% as a moderate clinical difference and, finally, a reduction in pain intensity ≥ 50% reflects substantial changes.

SECONDARY OUTCOMES:
Sleep quality | 4 weeks
  Pittsburgh Sleep Quality Index: designed by Buysse et al., it is a self-administered questionnaire that evaluates the quality and alterations of sleep in a one-month interval. Through nineteen individual items, scored from 0 "no difficulty" to 3 "severe difficulty", seven sleep components are assessed: 1) subjective quality of sleep, 2) sleep latency, 3) sleep duration, 4) efficiency usual sleep, 5) sleep disturbances, 6) use of medication for sleep and 7) daily functionality. The overall score can vary from 0 to 21 points, 0 indicating no difficulty and 21 severe difficulties in all areas. The Spanish version was validated in a sample of people diagnosed with FM showing a Cronbach's alpha coefficient of 0.805 and Spearman's correlation coefficient of 0.0773 (p <0.001) for the total score demonstrating a good internal consistency and an acceptable test-retest realiability.
Pain Catastrophizing | 4 weeks
  Pain Catastrophizing Scale: It is a self-administered questionnaire developed by Sullivan et al. in 1995 with the objective of measuring the impact of catastrophic thoughts on the experience of pain. The Pain Catastrophizing Scale comprises three dimensions of pain catastrophizing: 1) rumination 2) magnification and 3) helplessness which are assessed in 13 items.
  The Spanish version was validated in people diagnosed with FM by García-Campayo et al. with a sample of 230 participants in 2008. The results showed that the scale presented the same factorial structure of the three dimensions and showed adequate psychometric properties, with a Cronbach's alpha coefficient of 0.79 and an intraclass ratio of 0.84.
  A reduction of the 15-30% is established as the minimum clinically significant change, changes between 30 and 50% are moderately clinically significant and reductions of ≥50% are indicative of substantial clinical improvement.
Dysfunctional Beliefs and Attitudes about Sleep | 4 weeks
  Dysfunctional Beliefs and Attitudes about Sleep Scale: The original full version was created by Morin in 1994 to evaluate dysfunctional thoughts that cause and / or maintain insomnia. It consists of 30 items that are grouped into five theoretical dimensions: 1) consequences of insomnia on the state of mind, greeting or daily activity, 2) Concerns about loss of control and prediction of sleep, 3) Unrealistic expectations about the need for sleep, 4) Causal attributions of insomnia and 5) Beliefs about habits or behaviors that favor sleep.
Health status and quality of life associated with fibromyalgia | 4 weeks
  The Revised Fibromyalgia Impact Questionnaire (FIQ-R): developed by Bennet et al. in 2009 and validated into Spanish by Salgueiro et al. in 2013. This is the most current version of the Fibromyalgia Impact Questionnaire that was created and validated in 1991 by Burkhardt, Clark & Bennet. The FIQ-R is a self-administered questionnaire consisting of 21 items that are analog visual scales with eleven boxes that establish a score from 0 to 10.
  The maximum total score of the questionnaire is 100 and results from the sum of the scores of the three parameters described, representing the total impact of the symptoms on the quality of life.
  The minimum clinically significant change for the FIQ-R is a total score change of 27.04 point or a 45.5% change.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Climent Sanz, PhDc, Principal Investigator — Universitat de Lleida
Locations (1):
- Faculty of Nursing and Physiotherapy, University of Lleida, Lleida, Spain

REFERENCES:
- [Derived] Climent-Sanz C, Gea-Sanchez M, Moreno-Casbas MT, Blanco-Blanco J, Garcia-Martinez E, Valenzuela-Pascual F. A web-based therapeutic patient education intervention for pain and sleep for women with fibromyalgia: A sequential exploratory mixed-methods research protocol. J Adv Nurs. 2020 Jun;76(6):1425-1435. doi: 10.1111/jan.14333. Epub 2020 Mar 8. PMID 32068285